CLINICAL TRIAL: NCT03902665
Title: Up-front Hematopoietic Stem Cell Transplantation in Patients With Acute Myeloid Leukemia Aged 65-75
Brief Title: Up-front Hematopoietic Stem Cell Transplantation in Acute Myeloid Leukemia Patients Aged 65-75
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Principal Investigator, BACIGALUPO ANDREA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1749
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic hematopoietic stem cell transplantation (Experimental): Day -6, -5 Thiotepa 5 mg/kg/day . Day -4 to -3 Busulfan i. v 3,2 mg/kg/day and fludarabine i.v. 50 mg/m2 /day Day -2 fludarabine i.v. 50 mg/m2 Day -1 Rest Day 0 Begin cyclosporine; Infusion of T cell replete bone marrow transplant Day 1 Begin mycophenolate mofetil Day 3 and 5 Cyclophosphamide 50 mg/kg IV and Mesna Day 6 G-colony stimulating factor
  Interventions: Drug: Up-front allogeneic hematopoietic stem cell transplantation (HSCT)

INTERVENTIONS:
Drug: Up-front allogeneic hematopoietic stem cell transplantation (HSCT) — Patients classified as fit/unfit are included in the HSCT program. There are two early approaches allowed. A) Patients will be left untreated until HSCT B) Patients will receive 1 short course of chemotherapy before HSCT (Ara-C and anthracycline).
  Selection of strategy A or B, will be patient based on disease characteristics and dynamics or presence of high tumor load.
  Conditioning for haplo-HSCT should be started as soon as possible, within day 45 after initial diagnosis. This is to avoid delayed transplantation. Two dosing levels of the Thiotepa-Busulfan-Fludarabine (TBF) based protocol are allowed based on the clinical condition of the patient: fit patients below 70 will receive the TBF with 2 days of Busulfan, whereas patients with poorer clinical condition or above the age of 70 will receive a dose-reduced TBF, in which Busulfan may be reduced to 1 day only.
  Other Names: HSCT

SUMMARY:
Patients with acute myeloid leukemia aged 65-75 have a very poor prognosis, irrespective of the treatment strategy, including demethylating agents or conventional chemotherapy. With these approaches, remission rates do not exceed 40%, and overall disease-free survival at 1 year is in the order of 15%. The hypothesis is that up-front allogeneic hematopoietic stem cell transplant will produce a complete remission rate of 60% on day +56-70, and disease-free survival at 1 year of 30%. This is a single arm phase II study of upfront allogeneic stem cell transplantation, for patients with acute myeloid leukemia aged 65-75: the primary endpoint is a complete remission rate on day +56-70. The secondary endpoint is a 1-year overall disease-free survival of 30%.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65-75
* Patients with de novo or secondary acute myeloid leukemia (AML) - intermediate or high risk according to European LeukemiaNet (ELN) recommendations 2017
* Untreated patients at diagnosis of acute myeloid leukemia - patients may have received treatment for high-risk myelodysplastic syndromes with hypomethylating agents (HMA). They should not have received a course of induction chemotherapy to be eligible for this study
* Haploidentical family stem cell donor or other suitable donors available
* Fit and unfit patients by geriatric scale assessment
* Signed informed consent.

Exclusion Criteria:

* Acute Myeloid Leukemia good risk according to European LeukemiaNet 2017
* Positive serology for Human Immunodeficiency Virus.
* Serious organ dysfunction: left ventricular ejection fraction < 40%, forced expiratory volume in one second (FEV1), forced vital capacity (FVC) and diffusing capacity of the lung for carbon monoxide (DLCO) <50% of predicted, Liver Function Tests > 5 x the upper limit of normal, or creatinine clearance <30 ml/min .
* Life expectancy less than 30 days.
* Frail patients by geriatric scale assessment

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of complete remission equal or higher than 60% | From day 56 to day +70 post-transplant
  As a primary outcome measure, the rate of complete remission in treated patients will be evaluated. Complete remission will be assessed from days +56 to days +70 after transplant. A complete remission rate equal to or higher than 60% is expected.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bacigalupo, Prof., Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy